CLINICAL TRIAL: NCT01325701
Title: A Multicenter, Open-label, Phase 2, Safety and Efficacy Study of the Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI-32765, in Subjects With Relapsed or Refractory or de Novo Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Safety and Efficacy Study of a BTK Inhibitor in Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1106-CA; PCI-32765 (Other: Pharmacyclics)
Record Dates: First submitted 2011-02-02; First posted 2011-03-30 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Diffuse Large Cell B-lymphoma
Keywords: PCI-32765; Lymphoma, B-Cell; Bruton's Tyrosine Kinase; Non Hodgkin's Lymphoma; Germinal Center B-Cell; Activated B-Cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCI-32765: 560 mg (Experimental): Treatment Group 1: Subjects received 560 mg of ibrutinib once daily, on a continuous basis.
  Interventions: Drug: ibrutinib
- PCI-32765: 840 mg (Experimental): Treatment Group 2: Subjects received 840 mg of ibrutinib once daily, on a continuous basis.
  Interventions: Drug: ibrutinib

INTERVENTIONS:
Drug: ibrutinib — ibrutinib is an inhibitor of BTK
  Other Names: PCI-32765, Imbruvica

SUMMARY:
The purpose of this study is to evaluate the efficacy of ibrutinib (PCI-32765) in relapsed/refractory de novo activated B-cell (ABC) and germinal-cell B-Cell (GCB) Diffuse Large B-cell Lymphoma (DLBCL).

DETAILED DESCRIPTION:
The primary objectives of this study were to evaluate the efficacy of ibrutinib administered at 560 mg once per day in relapsed or refractory de novo ABC and GCB DLBCL, and to evaluate the efficacy of ibrutinib administered at 840 mg once per day in relapsed or refractory de novo ABC DLBCL.

The secondary objective was to evaluate the safety and tolerability of a fixed daily oral dosing regimen of ibrutinib in relapsed/refractory de novo DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. ECOG performance status ≤ 2.
3. Pathologically confirmed de novo DLBCL
4. Subjects must have available tissue for central pathology review to be eligible. Treatment Group 2: Subjects will be eligible if they have the non-GCB phenotype, as confirmed by Central IHC testing by the Hans method.
5. Relapsed or refractory disease, defined as either: 1) recurrence of disease after a CR, or 2) PR, SD, or progressive disease (PD) at completion of the treatment regimen preceding entry to the study (residual disease): Subjects must have previously received an appropriate first-line treatment regimen. Subjects who have not received HDT/ASCT must be ineligible for HDT/ASCT
6. Treatment Group 1: Subjects must have ≥ 1 measurable (> 2 cm in longest dimension) disease sites on CT scan. Treatment Group 2: Subjects must have ≥ 1 measurable (> 1.5 cm in longest dimension) disease sites on CT scan.

Exclusion Criteria:

1. Transformed DLBCL or DLBCL with coexistent histologies (eg, FL or MALT).
2. Primary mediastinal (thymic) large B-cell lymphoma.
3. Known central nervous system lymphoma. In addition, for subjects in Treatment Group 2, known leptomeningeal involvement is exclusionary.
4. Certain exclusions on prior therapy
5. Major surgery within 2 weeks of first dose of study drug.
6. Any of the following laboratory abnormalities:

   1. ANC < 0.75 x 10^9/L. Treatment Group 2: Eligible subjects must be independent of growth factor support for 7 days prior to the screening lab tests.
   2. Platelet count < 50 x 10^9/L independent of transfusion support. Treatment Group 2 only: Eligible subjects must be independent of transfusion support for 7 days prior to the screening lab tests.
   3. AST or ALT ≥ 3.0 x upper limit of normal (ULN)
   4. Creatinine > 2.0 x ULN
   5. Treatment Group 2 only: Hemoglobin < 8.0 g/dL
   6. Treatment Group 2 only: Total Bilirubin > 1.5 x ULN
7. Requires or has received anticoagulation treatment with warfarin or equivalent Vitamin K antagonists (eg, phenprocoumon)
8. Treatment Group 2: Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
9. Treatment Group 2: Known bleeding diathesis, eg, von Willebrand's disease, hemophilia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Beaupre, MD, Study Director — Pharmacyclics LLC.
Locations (15):
- United States (15):
  - UCLA Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - National Cancer Institute, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York University, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester School of Medicine and Dentistry, Rochester, New York
  - The Ohio Sate university, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Univerity of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson WH, Young RM, Schmitz R, Yang Y, Pittaluga S, Wright G, Lih CJ, Williams PM, Shaffer AL, Gerecitano J, de Vos S, Goy A, Kenkre VP, Barr PM, Blum KA, Shustov A, Advani R, Fowler NH, Vose JM, Elstrom RL, Habermann TM, Barrientos JC, McGreivy J, Fardis M, Chang BY, Clow F, Munneke B, Moussa D, Beaupre DM, Staudt LM. Targeting B cell receptor signaling with ibrutinib in diffuse large B cell lymphoma. Nat Med. 2015 Aug;21(8):922-6. doi: 10.1038/nm.3884. Epub 2015 Jul 20. PMID 26193343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 78 subjects were enrolled: 70 were treated with PCI-32765 (ibrutinib) 560 mg daily, and 8 were treated with ibrutinib 840mg daily. All subjects received at least 1 dose of study drug.
Period: Overall Study
Arm/Group | PCI-32765: 560 mg | PCI-32765: 840 mg
Started | 70 | 8
Completed | 49 | 5
Not Completed | 21 | 3
Not completed — Adverse Event | 12 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Rollerover Extension Study | 4 | 0

BASELINE CHARACTERISTICS:
Population: A total of 78 subjects were enrolled: 70 in PCI-32765: 560 mg , and 8 in PCI-32765: 840 mg . All subjects received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PCI-32765: 560 mg | PCI-32765: 840 mg | Total
Number analyzed (Participants) | 70 | 8 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 4 | 42
  >=65 years | 32 | 4 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (13.40) | 64.4 (13.96) | 62.7 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 2 | 22
  Male | 50 | 6 | 56
Region of Enrollment [Number; unit: participants]
  United States | 70 | 8 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Overall Response to Study Drug
Description: The primary endpoint of the study was overall response rate (ORR), defined as the proportion of participants who achieved a best overall response of complete response (CR) or partial response (PR), according to the revised International Working Group Criteria for non-Hodgkin's lymphoma (Cheson et al, 2007), as assessed by the investigator.
Time Frame: The median follow up time on the study for all treated participants is 1.7 months (range 0.1- 32.3 months)
Measure: Number; unit: percentage of participants
Arm/Group | PCI-32765: 560 mg | PCI-32765: 840 mg
Number analyzed (Participants) | 70 | 8
percentage of participants | 24.3 | 12.5

2. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Participants will be followed until progression of the disease or start of another anticancer treatment. The clinical database captured all AEs from baseline through end of treatment. Treatment Emergent AEs were collected pre-dose, at the beginning of each cycle and 30 days post last dose of study drug, unless related to study drug.
Time Frame: Adverse events determined to be related to study drug are collected from first dose until study exit (approximately 3 years).
Measure: Number; unit: participants
Arm/Group | PCI-32765: 560 mg | PCI-32765: 840 mg
Number analyzed (Participants) | 70 | 8
participants | 70 | 8

3. Secondary Outcome: Ibrutinib and Its Metabolite (PCI-45227) AUC0-24h After Repeat Dosing of PCI-32765
Description: Treatment Group 1 PK collection schedule:
  Cycle 1 Day 1: Pre-dose, 1, 2, 4, 7, and 24 hours post-dose Cycle 1 Day 8: Pre-dose, 1, 2, 4, 7, and 24 hours post-dose Cycle 1 Day 15: Pre-dose and 2 hours post-dose Cycle 1 Day 22: Pre-dose and 2 hours post-dose
  Treatment Group 2 PK collection schedule:
  Cycle 1 Day 8: Pre-dose, 1, 2, 4 and 7 hours post-dose Cycle 1 Day 15: Pre-dose and 2 hours post-dose Cycle 1 Day 22: Pre-dose and 2 hours post-dose Cycle 3 Day 1: Pre-dose, 1, 2, and 4 hours post-dose
Time Frame: Performed during the first month of receiving study drug.
Population: PK samples were collected in all participants (n=70 and 8 in PCI-32765: 560 mg and 840 mg, respectively). Of these, 59 participants in PCI-32765: 560 mg and 7 in PCI-32765: 840 mg on Cycle 1 Day 8 were evaluable for PK.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | PCI-32765: 560 mg | PCI-32765: 840 mg
Number analyzed (Participants) | 59 | 7
ng*h/mL
  PCI-32765 - Day 8 | 1285 (971) | 1337 (1556)
  PCI-45227 (Metabolite)- Day 8 | 1485 (948) | 1671 (1147)

ADVERSE EVENTS:
Arm/Group | PCI-32765: 560 mg | PCI-32765: 840 mg
Serious Adverse Events (participants affected / at risk) | 40/70 | 3/8
Other Adverse Events (participants affected / at risk) | 70/70 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765: 560 mg (N=70) | PCI-32765: 840 mg (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Localised oedema (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 1
Sepsis (Infections and infestations) | 3 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Brain mass (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765: 560 mg (N=70) | PCI-32765: 840 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 20 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 3 | 0
Eye pain (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 28 | 3
Nausea (Gastrointestinal disorders) | 24 | 4
Constipation (Gastrointestinal disorders) | 11 | 1
Vomiting (Gastrointestinal disorders) | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 4 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gingivitis ulcerative (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 30 | 0
Pyrexia (General disorders) | 14 | 1
Oedema peripheral (General disorders) | 12 | 1
Chills (General disorders) | 5 | 1
Pain (General disorders) | 5 | 1
Asthenia (General disorders) | 4 | 0
Local swelling (General disorders) | 4 | 0
Localised oedema (General disorders) | 3 | 0
Face oedema (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Catheter site erythema (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Suprapubic pain (General disorders) | 1 | 0
Tenderness (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 1
Urinary tract infection (Infections and infestations) | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 3 | 0
Candida infection (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 11 | 1
Alanine aminotransferase increased (Investigations) | 6 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 2
Lymphocyte count decreased (Investigations) | 8 | 0
Blood bilirubin increased (Investigations) | 6 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 1
International normalised ratio increased (Investigations) | 6 | 0
White blood cell count decreased (Investigations) | 6 | 0
Blood creatinine increased (Investigations) | 5 | 0
Neutrophil count decreased (Investigations) | 4 | 1
Weight decreased (Investigations) | 4 | 0
Weight increased (Investigations) | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0
Amylase increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 7 | 2
Headache (Nervous system disorders) | 7 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Brain mass (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 3
Anxiety (Psychiatric disorders) | 5 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 1
Jugular vein distension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
PCI-32765:840 mg:8 subjects were enrolled and followed through their 1st response assessment. Due to a lack of positive responses observed, enrollment was terminated for futility. Response rate should not be generalized due to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No